CLINICAL TRIAL: NCT00216125
Title: A Phase III Trial of Cisplatin/Etoposide/Radiotherapy With or Without Consolidation Docetaxel in Patients With Inoperable Locally Advanced Stage III Non-Small Cell Lung Cancer (NSCLC): Hoosier Oncology Group LUN01-24
Brief Title: Cisplatin/Etoposide/Radiotherapy +/- Consolidation Docetaxel in Advanced Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nasser Hanna, M.D. (Other)
Collaborators: Sanofi (Industry); Walther Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Nasser Hanna, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HOG LUN01-24
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Radiation; Docetaxel; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pre-Randomization (Other): Prior to randomization patients received Cisplatin 50 mg/m^2 days 1,8,29,36 + Etoposide 50 mg/m^2 days 1-5, 29-33 + Radiation 5940 cGy (180 cGy/day). Patients with CR, PR or SD with manageable toxicity were randomized to either Docetaxel arm or Observation only arm.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Radiation: Radiation
- Consolidation Docetaxel (Active Comparator): Docetaxel 75 mg/m^2 q3wk X 3 cycles.
  Interventions: Drug: Docetaxel
- Observation Only (No Intervention): Patients were followed for Observation.

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 50 mg/m2 day 1, 8, 29, 36
  Other Names: Platinol
  Arms: Pre-Randomization
Drug: Etoposide — Etoposide 50 mg/m2, days 1-5, 29-33
  Other Names: VP-16
  Arms: Pre-Randomization
Radiation: Radiation — Radiation 5940 cGy (180 cGy/day)
  Arms: Pre-Randomization
Drug: Docetaxel — docetaxel 75mg/m2 q3wk x 3 cycles
  Other Names: Taxol
  Arms: Consolidation Docetaxel

SUMMARY:
In a previous phase II study, patients with pathological stage IIIb (without pleural effusion) NSCLC were treated with concurrent cisplatin and etoposide plus thoracic radiotherapy followed by 3 cycles of consolidation therapy with docetaxel. Docetaxel was selected based upon a survival benefit in patients with recurrent NSCLC.

This trial will evaluate the role of consolidation therapy with docetaxel in patients with unresectable stage III disease. The purpose of the trial is to evaluate survival and toxicities of the regimens employed.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Cisplatin 50 mg/m2 d1, 8, 29, 36
* Etoposide 50 mg/m2/day d1-5, 29-33
* Radiation 5940 cGy (180 cGy/day)

Patients with CR, PR, SD Randomized to either:Docetaxel75 mg/m2 q3wk X 3 cycles

or Observation Only

Performance Status: ECOG 0 or 1

Life Expectancy: Not specified

Hematopoietic:

* ANC > 1,500/mm3
* Platelet count > 100,000/mm3
* Hemoglobin > 8 g/dl. PRBC transfusions will be allowed to increase hemoglobin to >8 g/dl

Hepatic:

* Serum bilirubin < institutional upper limit of normal (ULN)
* AST < 2.5 X the upper limits of normal if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 4 X ULN if AST are < ULN

Renal:

* Serum creatinine of < 2 mg/dl or calculated creatinine clearance > 50 cc/min

Cardiovascular:

* No clinically significant history of cardiac disease, (i.e. uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the past year, or cardiac ventricular arrhythmias requiring medication).

Pulmonary:

* Pre-registration FEV1 > 1 liters by spirometry within 42 days prior to study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic evidence of NSCLCUnresectable Stage IIIA (N2) OR Stage IIIB NSCLC.
* Unresectable Stage IIIA will be defined by the following criteria:
* N2 mediastinal lymph nodes must be multiple and/or bulky on CT scan such that in the opinion of the treating investigator, the patient is not a candidate for surgical resection
* N2 disease must be documented by biopsy, FDG-PET scan imaging, or by CT if nodes are > 2 cm on CT scan
* Stage IIIb patients must have N3 or T4 status. N3 status must be documented by one of the following criteria:
* Contralateral (to the primary tumor) mediastinal lymph node, supraclavicular or scalene lymph nodes proven by biopsy, FDG-PET scan imaging, or by CT if nodes are > 2 cm on CT scan.
* Patients with positive supraclavicular or scalene lymph nodes must not have disease extending up into the cervical region.
* All patients must have measurable or evaluable disease documented by CT, MRI, X-ray or physical exam within 28 days prior to study treatment.
* Negative pregnancy test

Eligibility for Consolidation Therapy

* Following completion of induction chemoradiotherapy patients without local progression of disease or distant metastases will then be randomized to receive consolidation therapy with docetaxel or observation. Patients will be stratified and randomized based on stage IIIa vs IIIb disease at baseline, CR vs. non-CR following induction chemoradiation, and ECOG PS 0 or 1 vs. 2.
* Patients must have completed chemoradiotherapy per protocol and at least 4 weeks but no more than 8 weeks must have elapsed from the last day of induction therapy (the last day of radiation) to be eligible for randomization to consolidation with docetaxel or observation.
* Patients must have undergone re-staging tests according to the study calendar and determined to have no evidence of disease progression to be eligible for randomization to consolidation with docetaxel or observation.
* Patients must have an ANC > 1,500/mm3, platelet count > 100,000/ mm3, and hemoglobin > 8 g/dl obtained within 14 days prior to registration for randomization to consolidation with docetaxel or observation.
* Patients must have adequate hepatic function as defined by a serum bilirubin < institutional upper limit of normal (ULN) and an AST and/or ALT < 2.5 X the upper limits of normal if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 4 X ULN if transaminases are < ULN within 14 days prior to registration for randomization to consolidation with docetaxel or observation.

Exclusion Criteria:

* No prior chemotherapy or radiotherapy for lung cancer.
* No unintended weight loss > 5% body weight in the preceding 3 months prior to study treatment will not be eligible for this trial.
* No symptomatic peripheral neuropathy prior to entry onto the study. Peripheral neuropathy must be < Grade 1 to be eligible.
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years.
* No history of allergic reactions to drugs utilizing the vehicle polysorbate 80 (docetaxel) and polysorbate 80 + polyethylene glycol (etoposide).
* If the patient has hearing loss at pre-study, performance of an audiogram is recommended (not mandatory) to document baseline hearing status in the event of possible further hearing loss due to cisplatin administration.
* No current breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2002-02; Primary Completion 2006-06 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (15):
- United States (15):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - AP&S Clinic, Terre Haute, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Methodist Cancer Center, Omaha, Nebraska
  - US Oncology, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hanna N, Neubauer M, Yiannoutsos C, McGarry R, Arseneau J, Ansari R, Reynolds C, Govindan R, Melnyk A, Fisher W, Richards D, Bruetman D, Anderson T, Chowhan N, Nattam S, Mantravadi P, Johnson C, Breen T, White A, Einhorn L; Hoosier Oncology Group; US Oncology. Phase III study of cisplatin, etoposide, and concurrent chest radiation with or without consolidation docetaxel in patients with inoperable stage III non-small-cell lung cancer: the Hoosier Oncology Group and U.S. Oncology. J Clin Oncol. 2008 Dec 10;26(35):5755-60. doi: 10.1200/JCO.2008.17.7840. Epub 2008 Nov 10. PMID 19001323
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 77 patients who started the pre-randomization arm were not randomized due to the following reasons: toxicities, disease progression, ineligibility, patient decision, death, physician decision, and other miscellaneous reasons. Only patients who were randomized to consolidation therapy or observation are included in the study analysis.
Period: Pre-Randomization Phase
Arm/Group | Pre-Randomization | Consolidation Docetaxel | Observation Only
Started | 243 | 0 | 0
DSMB Cohort for Futility | 203 | 0 | 0
Completed | 166 | 0 | 0
Not Completed | 77 | 0 | 0
Period: Randomization Phase
Arm/Group | Pre-Randomization | Consolidation Docetaxel | Observation Only
Started | 0 | 84 | 82
DSMB Cohort for Futility | 0 | 73 | 74
Completed | 0 | 73 | 74
Not Completed | 0 | 11 | 8

BASELINE CHARACTERISTICS:
Arm/Group | Pre-Randomization
Number analyzed (Participants) | 243
Age, Continuous [Median (Standard Deviation); unit: years] | 63.0 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 161
Region of Enrollment [Number; unit: participants]
  United States | 243
Percentage of participants with Stage IIIa vs IIIb disease at baseline [Number; unit: percentage] | 41.15

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: A comparison of overall survival following cisplatin/etoposide/radiotherapy between the consolidation docetaxel and observation arms was analyzed using Kaplan-Meier analysis. Median survival time and a log rank test were used to analyze the hypothesized improvement in overall survival.
Time Frame: Participants were measured from treatment initiation to death
Population: The analysis cohort for the results reported below are based on a planned interim DSMB evaluation conducted in 2006. This evaluation concluded that further accrual was futile and the study should be terminated. The 203 subjects included in this analysis had data sufficiently mature at the time of the DSMB analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Consolidation Docetaxel | Observation Only
Number analyzed (Participants) | 73 | 74
Months | 21.5 [17.0 to 34.8] | 24.1 [18.0 to 34.2]
Statistical Analysis 1: Comparison: Consolidation Docetaxel vs Observation Only; Test type: Superiority or Other; p = 0.883, Log Rank; Median Difference (Final Values) = 10

2. Secondary Outcome: Progression Free Survival
Description: A comparison of progression free survival following cisplatin/etoposide/radiotherapy between the consolidation docetaxel and observation arms was analyzed using Kaplan-Meier analysis. Median PFS time and a log rank test were used to analyze the hypothesized improvement in progression free survival.
  Progression is defined by RECIST as a 20% increase in the sum of longest diameters of target measurable lesions over the smallest sum observed (over baseline if no decrease during therapy) or by the appearance of a new lesion.
Time Frame: Participants were monitored from treatment initiation until disease progression per RECIST or death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Consolidation Docetaxel | Observation Only
Number analyzed (Participants) | 73 | 74
months | 12.3 [9.4 to 16.9] | 12.9 [8.3 to 17.1]

ADVERSE EVENTS:
Groups:
- Pre-Randomization: Prior to randomization patients received Cisplatin 50 mg/m^2 days 1,8,29,36 + Etoposide 50 mg/m^2 days 1-5, 29-33 + Radiation 5940 cGy (180 cGy/day). Patients with CR, PR or SD with manageable toxicity were randomized to either Docetaxel arm or Observation only arm.
  Cisplatin: Cisplatin 50 mg/m2 day 1, 8, 29, 36
  Etoposide: Etoposide 50 mg/m2, days 1-5, 29-33
  Radiation: Radiation 5940 cGy (180 cGy/day)
  Adverse events reported in this arm consist only of participants that were not randomized into the "Consolidation Docetaxel" or "Observation Only" arms.
Arm/Group | Pre-Randomization | Consolidation Docetaxel | Observation Only
Serious Adverse Events (participants affected / at risk) | 44/77 | 43/84 | 29/82
Other Adverse Events (participants affected / at risk) | 63/77 | 73/84 | 79/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Randomization (N=77) | Consolidation Docetaxel (N=84) | Observation Only (N=82)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
ANOREXIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
BLOOD/BONE MARROW - OTHER (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARRHYTHMIA - OTHER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC GENERAL - OTHER (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
CNS CEREBROVASCULAR ISCHEMIA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CONSTITUTIONAL SYMPTOMS - OTHER (General disorders) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Gastrointestinal disorders) | 5 (7) | 4 (5) | 6 (6)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 4 (4)
ESOPHAGITIS (Gastrointestinal disorders) | 7 (7) | 5 (5) | 8 (10)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 1 (1) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 8 (9) | 13 (15) | 4 (5)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1) | 1 (1) | 1 (1)
FISTULA, GI (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 1 (1) | 0 (0) | 0 (0)
HEMOGLOBIN (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4)
HEMORRHAGE, CNS (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
HEMORRHAGE, GI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
HEMORRHAGE/BLEEDING - OTHER (General disorders) | 1 (1) | 2 (2) | 0 (0)
HYPERTENSION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
INFECTION - OTHER (Infections and infestations) | 8 (9) | 11 (13) | 5 (5)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2)
METABOLIC/LABORATORY - OTHER (Investigations) | 1 (1) | 0 (0) | 0 (0)
MOOD ALTERATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (4) | 5 (6) | 0 (0)
NEUROLOGY - OTHER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 6 (6) | 3 (3) | 3 (3)
PAIN (General disorders) | 2 (2) | 2 (2) | 2 (2)
PAIN - OTHER (General disorders) | 2 (2) | 1 (1) | 1 (1)
PERICARDIAL EFFUSION (NON-MALIGNANT) (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 1 (1) | 1 (4) | 0 (0)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 0 (0) | 0 (0) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (1) | 1 (1) | 0 (0)
SOMNOLENCE/DEPRESSED LEVEL OF CONSCIOUSNESS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
SYNCOPE (FAINTING) (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 3 (3) | 3 (3) | 5 (5)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (5) | 5 (6) | 0 (0)
WEIGHT LOSS (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Randomization (N=77) | Consolidation Docetaxel (N=84) | Observation Only (N=82)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 1 (1) | 7 (9) | 1 (1)
ALKALINE PHOSPHATASE (Investigations) | 1 (1) | 6 (7) | 4 (4)
ALKALOSIS (METABOLIC OR RESPIRATORY) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 0 (0) | 2 (2) | 1 (1)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 0 (0) | 2 (2) | 4 (4)
ALLERGY/IMMUNOLOGY - OTHER (SPECIFY, __) (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 4 (4) | 1 (1) | 0 (0)
ANOREXIA (Gastrointestinal disorders) | 21 (31) | 27 (40) | 31 (41)
APNEA (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2) | 1 (2)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 2 (2) | 1 (1) | 1 (1)
AUDITORY/EAR - OTHER (SPECIFY, __) (Ear and labyrinth disorders) | 2 (2) | 5 (8) | 3 (4)
BICARBONATE, SERUM-LOW (Investigations) | 0 (0) | 2 (3) | 0 (0)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 2 (2) | 1 (1) | 2 (2)
BLOOD/BONE MARROW - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0)
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Investigations) | 0 (0) | 1 (2) | 0 (0)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 3 (4) | 5 (8) | 2 (3)
CARDIAC ARRHYTHMIA - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1) | 1 (1) | 2 (3)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 8 (9) | 7 (9) | 12 (13)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 1 (1) | 4 (4) | 1 (1)
COAGULATION - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
CONFUSION (Nervous system disorders) | 3 (5) | 0 (0) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 8 (12) | 22 (30) | 25 (29)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 0 (0) | 3 (3) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 29 (41) | 37 (51)
CREATININE (Investigations) | 6 (14) | 4 (4) | 4 (6)
CUSHINGOID APPEARANCE (E.G., MOON FACE, BUFFALO HUMP, CENTRIPETAL OBESITY, CUTANEOUS STRIAE) (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Gastrointestinal disorders) | 11 (11) | 9 (20) | 10 (10)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 10 (13) | 20 (29) | 11 (12)
DIZZINESS (Nervous system disorders) | 5 (6) | 14 (19) | 8 (12)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 5 (7) | 1 (1) | 5 (8)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 34 (40) | 40 (52) | 31 (43)
ESOPHAGITIS (Gastrointestinal disorders) | 24 (36) | 36 (68) | 42 (52)
EXTRAPYRAMIDAL/INVOLUNTARY MOVEMENT/RESTLESSNESS (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 39 (70) | 43 (88) | 49 (85)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 0 (0) | 7 (7) | 2 (2)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 3 (3) | 10 (13) | 7 (9)
FISTULA, GI (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FLUSHING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 2 (4) | 9 (13) | 6 (6)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 5 (11) | 10 (26) | 5 (9)
GLUCOSE, SERUM-LOW (HYPOGLYCEMIA) (Investigations) | 1 (1) | 1 (1) | 0 (0)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 21 (26) | 29 (37) | 35 (47)
HEARING: PATIENTS WITHOUT BASELINE AUDIOGRAM AND NOT ENROLLED IN A MONITORING PROGRAM (Ear and labyrinth disorders) | 0 (0) | 1 (3) | 4 (6)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 10 (12) | 13 (17) | 17 (24)
HEMOGLOBIN (Blood and lymphatic system disorders) | 20 (39) | 30 (62) | 26 (39)
HEMOGLOBINURIA (Investigations) | 0 (0) | 0 (0) | 1 (1)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 2 (2)
HEMORRHAGE, GI (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 8 (8) | 3 (3)
HEMORRHAGE/BLEEDING - OTHER (SPECIFY, __) (General disorders) | 2 (2) | 2 (2) | 1 (2)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 0 (0)
HOT FLASHES/FLUSHES (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERTENSION (Cardiac disorders) | 2 (2) | 3 (3) | 3 (3)
HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
HYPOTENSION (Cardiac disorders) | 7 (11) | 9 (10) | 3 (5)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 9 (13) | 15 (27) | 11 (17)
INFECTION WITH UNKNOWN ANC (Infections and infestations) | 2 (2) | 1 (3) | 1 (1)
INJECTION SITE REACTION/EXTRAVASATION CHANGES (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3)
INR (INTERNATIONAL NORMALIZED RATIO OF PROTHROMBIN TIME) (Surgical and medical procedures) | 0 (0) | 1 (5) | 0 (0)
INSOMNIA (General disorders) | 11 (14) | 11 (13) | 19 (25)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 26 (54) | 45 (114) | 34 (63)
LYMPHATICS - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 (7) | 8 (35) | 3 (6)
MAGNESIUM, SERUM-HIGH (HYPERMAGNESEMIA) (Investigations) | 1 (1) | 0 (0) | 0 (0)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 3 (3) | 3 (9) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
METABOLIC/LABORATORY - OTHER (SPECIFY, __) (Investigations) | 3 (4) | 5 (21) | 6 (14)
MOOD ALTERATION (Psychiatric disorders) | 7 (11) | 16 (21) | 18 (28)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) (Gastrointestinal disorders) | 11 (12) | 7 (16) | 8 (8)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (8) | 3 (5)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (SPECIFY, __) (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 1 (1)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 29 (44) | 32 (51) | 41 (67)
NEUROLOGY - OTHER (SPECIFY, __) (Nervous system disorders) | 4 (5) | 0 (0) | 0 (0)
NEUROPATHY: MOTOR (Nervous system disorders) | 3 (3) | 3 (5) | 2 (3)
NEUROPATHY: SENSORY (Nervous system disorders) | 7 (9) | 15 (19) | 15 (22)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 25 (38) | 50 (102) | 37 (62)
OCULAR/VISUAL - OTHER (SPECIFY, __) (Eye disorders) | 1 (1) | 1 (2) | 1 (1)
PAIN (General disorders) | 19 (28) | 28 (60) | 28 (53)
PAIN - OTHER (SPECIFY, __) (General disorders) | 23 (41) | 26 (39) | 29 (56)
PANCREATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (NON-MALIGNANT) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PHLEBITIS (INCLUDING SUPERFICIAL THROMBOSIS) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
PHOTOSENSITIVITY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PLATELETS (Blood and lymphatic system disorders) | 15 (31) | 24 (46) | 20 (34)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 1 (1)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 13 (17) | 4 (5)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 1 (1) | 3 (4) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 7 (8) | 5 (12) | 4 (6)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
PULMONARY FIBROSIS (RADIOGRAPHIC CHANGES) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (11) | 5 (12)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (10) | 7 (9)
RASH: DERMATITIS ASSOCIATED WITH RADIATION (Skin and subcutaneous tissue disorders) | 10 (11) | 8 (12) | 12 (18)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4)
RENAL/GENITOURINARY - OTHER (SPECIFY, __) (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
RIGORS/CHILLS (General disorders) | 2 (2) | 3 (3) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SODIUM, SERUM-HIGH (HYPERNATREMIA) (Investigations) | 0 (0) | 1 (4) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 4 (6) | 6 (9) | 5 (7)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA (Cardiac disorders) | 1 (1) | 5 (5) | 1 (1)
SWEATING (DIAPHORESIS) (General disorders) | 1 (1) | 6 (7) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 0 (0) | 5 (8) | 0 (0)
SYNDROMES - OTHER (SPECIFY, __) (General disorders) | 0 (0) | 1 (1) | 0 (0)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 2 (3) | 1 (1) | 1 (1)
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
THYROID FUNCTION, LOW (HYPOTHYROIDISM) (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
URIC ACID, SERUM-HIGH (HYPERURICEMIA) (Investigations) | 1 (1) | 1 (2) | 0 (0)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
VISION-BLURRED VISION (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 2 (2)
VOMITING (Gastrointestinal disorders) | 15 (19) | 22 (24) | 15 (23)
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
WEIGHT GAIN (General disorders) | 1 (1) | 1 (1) | 1 (2)
WEIGHT LOSS (General disorders) | 8 (9) | 15 (20) | 12 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No